CLINICAL TRIAL: NCT03208127
Title: Pan-genotypic Direct Acting Antiviral Therapy in Donor HCV-positive to Recipient HCV-negative Liver Transplant
Brief Title: DAA Treatment in Donor HCV-positive to Recipient HCV-negative Liver Transplant
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Protocol transitioned to standard of care, no funding available to continue support of research work or data analysis
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Raymond Chung, Director of Hepatology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017P000653
Record Dates: First submitted 2017-07-03; First posted 2017-07-05 (Actual); Results first posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: End Stage Liver Disease; Hepatitis C
Keywords: HCV; Epclusa; ESLD
MeSH Terms: conditions — End Stage Liver Disease; Hepatitis C | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with Direct Acting Antiviral (DAA) Fixed Dose Combination (Experimental): 12 weeks of HCV treatment with medically appropriate direct acting antiviral
  Interventions: Drug: Treatment with Direct Acting Antiviral tablet

INTERVENTIONS:
Drug: Treatment with Direct Acting Antiviral tablet — HCV Treatment for 12 Weeks
  Other Names: DAA

SUMMARY:
This is a single center study for the donation of Hepatitis C Virus (HCV)-positive livers to HCV negative recipient patients, with preemptive, interventional treatment to prevent HCV transmission upon transplantation.

DETAILED DESCRIPTION:
Patients will be selected based on diminished likelihood of receiving a liver from the waitlist within a period during which they would be likely to succumb to severe comorbidities. This will be determined in part through use of a patient's Model of End Stage Liver Disease (MELD) score, listing status, and clinical judgment. To ensure maximal benefit for the recipient, only high quality donor livers will be accepted.

ELIGIBILITY:
Inclusion Criteria:

* Recipient is Age ≥ 18 years
* Met Massachusetts General Hospital (MGH) transplant center criteria, listed for liver transplant
* HCV naïve
* Able to sign informed consent

Exclusion Criteria:

* Pregnant or nursing (lactating) women
* Human immunodeficiency virus (HIV) positivity
* Need for dual organ transplant
* Any contra-indication to liver transplantation per center protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Chung, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Masschusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Coded data is anticipated to be shared with potential collaborators.
Supporting Information: Study Protocol
Time Frame: Anticipated that data from the study will become available within 6 months after the final patient completes the primary study endpoint (12 weeks post treatment)
Access Criteria: Data would only be shared with Institutional Review Board (IRB) approved collaborators.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between November 2017 and March 2021. 33 subjects underwent liver transplant from an Hepatitis C Virus (HCV) Antibody (Ab) positive donor. 9 subjects received HCV Ab positive/HCV Ribonucleic acid (RNA) (Nucleic Acid Testing (NAT)-) donors and did not receive Direct Acting Antiviral (DAA) treatment. 24 subjects initiated treatment with DAAs.
Pre-assignment Details: Enrolled subjects who did not require treatment with direct acting antivirals were excluded from analysis.
Groups:
- Treatment With Direct Acting Antiviral Fixed Dose Combination: 12 weeks of HCV treatment with medically appropriate direct acting antiviral
  Treatment with Direct Acting Antiviral tablet: HCV Treatment for 12 Weeks
Period: Overall Study
Arm/Group | Treatment With Direct Acting Antiviral Fixed Dose Combination
Started | 24
Completed | 23
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Baseline Analysis population is number of consented subjects initiating Direct Antiviral Treatment
Arm/Group | Treatment With Direct Acting Antiviral Fixed Dose Combination
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 24
Recipient Negative HCV status at time of transplant [Count of Participants; unit: Participants] | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Undetectable Hepatitis C Virus (HCV) Viral RNA
Description: Number of dosed subjects with negative HCV viral RNA at 12 weeks after the last dose of treatment.
Time Frame: 12 weeks post treatment
Population: 1 subject died and was not included in analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Direct Acting Antiviral Fixed Dose Combination
Number analyzed (Participants) | 23
Participants | 23

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events and Out of Range Lab Values
Description: Safety and tolerability of direct acting antiviral therapy in the liver transplant patient will be monitored by quantifying the number of treatment related adverse events per patient and evaluating clinically significant out of range laboratory results as compared to baseline/pretreatment values per patient.
Time Frame: 12 weeks
Population: Number of participants receiving at least 1 dose of DAA treatment were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Direct Acting Antiviral Fixed Dose Combination
Number analyzed (Participants) | 24
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collect from time of Direct Acting Antiviral Treatment initiation through last dose of therapy, an average of 12 weeks.
Description: Only treatment emergent adverse events were collected.
Arm/Group | Treatment With Direct Acting Antiviral Fixed Dose Combination
All-Cause Mortality (participants affected / at risk) | 2/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

LIMITATIONS AND CAVEATS:
Protocol transitioned out of research to standard of care and was closed prior to completion and planned enrollment goal was not met. Review of data from enrolled patient was used for reporting purposes and data is primarily descriptive and not based on statistical analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/27/NCT03208127/Prot_SAP_000.pdf